CLINICAL TRIAL: NCT05084248
Title: Vitamin D Deficiency in Adults Following a Major Burn Injury
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Principal Investigator, Karen Kowalske, Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU-2019-1223
Record Dates: First submitted 2021-09-27; First posted 2021-10-19 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Vitamin D Deficiency; Burns
MeSH Terms: conditions — Vitamin D Deficiency; Burns | interventions — Ergocalciferols; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Low-dose (Active Comparator): 400 IU Per Orem
  Interventions: Drug: Ergocalciferol Capsules
- High-dose (Experimental): 4000 IU Per Orem
  Interventions: Drug: Ergocalciferol Capsules

INTERVENTIONS:
Drug: Ergocalciferol Capsules — Capsules of ergocalciferol at 400 IU and 4000 IU
  Other Names: Vitamin D

SUMMARY:
This is a single site double blind randomized controlled trial of replacing Vitamin D for Vitamin D-deficient burn patients at a current recommended dose (400 IU daily) versus a higher dose (4000 IU daily). Capsules will be made in a compounding pharmacy and will look identical.

Randomized controlled trial. People who meet the selection criteria will be randomized to either low or high dosage of Vitamin D. Treatment arm is high dose Vitamin D (4000 IU), and control is low dose Vitamin D (400 IU). Main outcome variables include PROMIS-29 measures of physical health, mental health and social health, the Veterans RAND 12 Item Health Survey (VR-12), and the 4-D Itch Scale. Secondary outcome variables include subject demographics, injury demographics and characteristics.

ELIGIBILITY:
Inclusion Criteria:

1. Adults, 18 years of age or older, who have completed 6 months from time of their burn injury
2. ≥ 10% TBSA, ≥ 65 years of age and Burn Surgery for Wound Closure
3. ≥ 20% TBSA, 18 - 64 of age and Burn Surgery for Wound Closure
4. Electrical high voltage / lightning and Burn Surgery for Wound Closure
5. Hand burn and/or face burn, and/or feet burn and Burn Surgery for Wound Closure
6. May speak English or Spanish
7. Vit. D deficiency

Exclusion Criteria:

1. Patients with parathyroid disease, severe liver dysfunction, sever kidney dysfunction, which are not caused by the burn injury
2. Patients with malignant tumors
3. Patients not meeting the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-09-29 (Actual); Primary Completion 2025-08-18 (Actual); Study Completion 2025-08-18 (Actual)

PRIMARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System-29 | 6 months and 12 months
  Measures change in physical health, mental health and social health between time points.
  When the scores are transformed into t-score metric, all PROMIS measures range from 0-100. For each domain, the higher scores indicate more of what is being measured. Therefore, higher scores on anxiety indicate more anxiety, while higher scores on physical function indicate higher physical function. Please see more information here: https://www.healthmeasures.net/explore-measurement-systems/promis/intro-to-promis.

SECONDARY OUTCOMES:
Demographics | 6 months
  include subject demographics, injury demographics and characteristics
Patient-Reported Outcomes Measurement Information System-Global | 6 months and 12 months
  Measures change in emotional, physical, and social health between timepoints.
  When the scores are transformed into t-score metric, all PROMIS measures range from 0-100. For each domain, the higher scores indicate more of what is being measured. Therefore, higher scores indicates a higher global health.
Patient-Reported Outcomes Measurement Information System-Itch | 6 months and 12 months
  Measures change in itch between timepoints. When the scores are transformed into t-score metric, all PROMIS measures range from 0-100. For each domain, the higher scores indicate more of what is being measured. Therefore, higher scores indicate more itch.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Pia Kabamalan, Study Chair — UT Southwestern
Locations (1):
- Parkland Health and Hospital Systems, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data may be shared with Burn Model System under National Institute on Disability and Rehabilitation Research.

DOCUMENTS (1):
  • Informed Consent Form (2022-10-19): https://cdn.clinicaltrials.gov/large-docs/48/NCT05084248/ICF_000.pdf